CLINICAL TRIAL: NCT06015100
Title: Efficacy and Safety of Inetetamab Plus Pyrotiniband and Capecitabine in HER2-positive Metastatic Breast Cancer Patients With or Without Brain Metastasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yan Xue (Other)
Responsible Party: Sponsor-Investigator, Yan Xue, Director of tumor hospital, Xi'an International Medical Center Hospital
Organization: Xi'an International Medical Center Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORP-239-Ｎ3
Record Dates: First submitted 2023-08-08; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Label 1 (Experimental): Inetetamab plus pyrotiniband and capecitabine
  Interventions: Drug: Inetetamab plus pyrotiniband and capecitabine

INTERVENTIONS:
Drug: Inetetamab plus pyrotiniband and capecitabine — Inetetamab plus pyrotiniband and capecitabine

SUMMARY:
This study intends to include HER2-positive metastatic breast cancer patients (with or without brain metastasis) who have become resistant to previous treatment with trastuzumab. It will use pertuzumab in combination with pyrotinib and capecitabine to observe efficacy and safety. The choice of capecitabine as the chemotherapy drug is mainly based on the following reasons: ① it has been less commonly used as neoadjuvant treatment, making it less prone to cross-resistance; ② its oral formulation is convenient for administration, making it more acceptable to patients; ③ previous studies have shown good efficacy when combined with pyrotinib; ④ previous research in breast cancer patients with brain metastasis has also demonstrated certain effectiveness. It is hoped that through this study, preliminary evidence can be provided for the dual-target treatment of original Chinese drugs, as well as the treatment of HER2+ MBC after resistance to trastuzumab, and the addition of new data for patients with brain metastasis.

DETAILED DESCRIPTION:
Research Title A single-center, open-label, single-arm clinical study on the efficacy and safety of pertuzumab in combination with pyrotinib and capecitabine in the treatment of HER2-positive metastatic breast cancer patients who have developed resistance to previous trastuzumab treatment (with or without brain metastasis).

Study Drugs - Injectable pertuzumab: 50mg/vial - Pyrotinib: 80mg/tablet

Research Objective To evaluate the effectiveness and safety of pertuzumab in combination with pyrotinib and capecitabine in the treatment of HER2-positive metastatic breast cancer patients who have developed resistance to previous trastuzumab treatment (with or without brain metastasis). This study aims to provide preliminary evidence for the dual-target treatment of original Chinese drugs, and to add new data to the treatment model for trastuzumab-resistant HER2+ MBC and patients with brain metastasis.

Study Design A single-center, open-label, single-arm clinical study with a planned enrollment of 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can voluntarily sign an informed consent form;
* Females aged ≥18 years at the time of signing the informed consent form;
* ECOG PS performance status score between 0 and 2;
* Patients histologically diagnosed with HER2-positive metastatic breast cancer, with or without brain metastasis, and with locally recurrent disease that cannot undergo curative surgery or radiation therapy;
* Patients who experience relapse or metastasis within 1 year during or after (neo)adjuvant pertuzumab-based targeted therapy, or disease progression during first-line pertuzumab-based targeted therapy in advanced stages;
* Patients who have received ≤1 regimen of previous pertuzumab-based targeted therapy for recurrent or metastatic disease;
* Brain metastasis patients must meet the following criteria: stable previous brain metastasis treatment, untreated brain metastasis with no immediate need for local treatment, or progressive previous brain metastasis without immediate need for local treatment;
* Left ventricular ejection fraction (LVEF) ≥50%;
* Blood routine examination meets the following conditions: ① absolute neutrophil count (ANC) ≥1.5×109/L, ② platelet count ≥100×109/L, ③ hemoglobin ≥90g/L, ④ white blood cell count ≥3.0×109/L;
* Liver function meets the following conditions: ① serum total bilirubin ≤1.5×ULN, or ≤3×ULN if liver metastasis is present, ② aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤3×ULN, or ≤5×ULN if liver metastasis is present;
* Renal function meets the following conditions: serum creatinine ≤1.5×ULN or creatinine clearance ≥50 mL/min (creatinine clearance calculated according to the Cockcroft-Gault formula);
* Female patients who meet the following conditions can participate in this study: ① not fertile; ② fertility potential, with a negative pregnancy test result within 7 days before the first administration of the study drug, not breastfeeding, and consistently using highly effective contraceptive measures before study enrollment, throughout the study period, and within 6 months after the last administration of the study drug.

Exclusion Criteria:

* Those who have previously received Inetetamab and/or pyrotinib treatment;
* Those who have received capecitabine treatment within the past 2 weeks before randomization;
* Patients with noticeable symptoms who require immediate local treatment for brain metastasis;
* Exclusion criteria include having had or currently having any other malignant tumors within the past 5 years, except for cured cervical intraepithelial neoplasia, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (in situ carcinoma), and T1 (tumor invasion of the basement membrane)];
* Exclusion criteria include having undergone major surgical procedures (including thoracotomy biopsy) within the past 4 weeks before randomization, suffering from major trauma (such as bone fracture), having unhealed wounds or fractures at the time of screening, or anticipating the need for major surgery during the study treatment period;
* Exclusion criteria include having a history of myocardial infarction within the past 6 months; New York Heart Association (NYHA) class ≥ II congestive heart failure history, severe arrhythmia uncontrolled by medication (excluding atrial fibrillation, paroxysmal supraventricular tachycardia); known decrease in left ventricular ejection fraction (LVEF) to below 50% during or after previous trastuzumab treatment;
* Known allergy to the drugs and excipients involved in this trial;
* Known history of hypersensitivity reactions to any investigational drug;
* Subjects deemed unfit for participation by other researchers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-20 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  It is an indicator of the long-term efficacy of the drug

SECONDARY OUTCOMES:
Objective Response Rate | 4 weeks
  The proportion of patients with the best response of complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST).
Disease Control Rate | 4 weeks
  The proportion of patients with tumor shrinkage or stability maintained for a certain period, including cases of CR, PR, and stable disease (SD).
Overall survival | the time from randomization to death from any cause, assessed up to 100 months.
  It is an indicator of the long-term efficacy of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Yan Xue, Principal Investigator — Xi'an International Medical Center Hospital
Locations (1):
- Xi'an International Medical Center Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No